CLINICAL TRIAL: NCT00213551
Title: Comparative Effects of Glutamine and Glucose on Intestinal Protein Metabolism in Healthy Humans
Brief Title: Glutamine and Intestinal Protein Metabolism
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2003/037/HP
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2013-06-18 (Estimated); Status verified 2013-06

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Glutamine; Glucose

INTERVENTIONS:
Drug: Glutamine
Drug: Glucose
Drug: glutamine-antioxidants containing solution

SUMMARY:
Gut barrier plays a major role in defence of the organism. During catabolic states, like major surgery or inflammation, gut barrier could be altered. It has been reported that preoperative nutritional support may have beneficial effects on clinical outcome in patients with surgery on gastrointestinal tract. Glutamine, which is a conditionally essential amino, have been reported to modulate inflammatory, antioxidant responses and protein metabolism in intestine. In addition, glutamine supply improves clinical outcome in critically ill patients. Antioxidant micronutrients may also have some beneficial effects in intestine by improving antioxidant response and might also regulate protein expression. Nevertheless, effects of glutamine combined to antioxidant micronutrients have not been evaluated.

Thus, the aim of this study will be to assess the influence of glutamine and glutamine-antioxidant micronutrients-containing solutions on intestinal response in humans.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers, male and female, aged between 18 and 50 years, negatives for HIV1, 2 and for HVC and HVB
* BMI between 20 and 24 kg/m²,
* giving their written informed consent
* no-smokers
* no allergic and digestive antecedents

Exclusion Criteria:

* smokers
* Allergic and digestive antecedents,
* pregnancy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2004-04; Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Impact on protein synthesis rate and proteolytic activities in intestine. | at the end of infusion (hour 5)

SECONDARY OUTCOMES:
Comparison of protein expression pattern and glutathione synthesis. | at the end of infusion (hour 5)

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Déchelotte, MD, PhD, Principal Investigator — University Hospital, Rouen
Locations (1):
- University Hospital of Rouen, Rouen, France

REFERENCES:
- [Derived] Goichon A, Coeffier M, Claeyssens S, Lecleire S, Cailleux AF, Bole-Feysot C, Chan P, Donnadieu N, Lerebours E, Lavoinne A, Boyer O, Vaudry D, Dechelotte P. Effects of an enteral glucose supply on protein synthesis, proteolytic pathways, and proteome in human duodenal mucosa. Am J Clin Nutr. 2011 Sep;94(3):784-94. doi: 10.3945/ajcn.110.009738. Epub 2011 Jul 27. PMID 21795435